CLINICAL TRIAL: NCT01149915
Title: A Phase I Open-Label Study to Assess the Safety, Tolerability and Preliminary Efficacy of TH-302, a Hypoxia-Activated Prodrug, in Patients With Advanced Leukemias
Brief Title: Study of Hypoxia-Activated Prodrug TH-302 to Treat Advanced Leukemias
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Threshold Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TH-CR-407
Record Dates: First submitted 2010-06-01; First posted 2010-06-24 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Acute Myelogenous Leukemia; Acute Lymphoblastic Leukemia; Chronic Myelogenous Leukemia; High-risk Myelodysplastic Syndrome; Chronic Lymphocytic Leukemia; Advanced Myelofibrosis
Keywords: Advanced Leukemias; Relapsed/Refractory Leukemias; AML; ALL; CML; MDS; CLL; MF; Evofosfamide
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia | interventions — TH 302

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: TH-302 — TH-302 will be administered as a 30-minute intravenous infusion daily for 5 days every 21 days. Patients who successfully complete a 3-week treatment cycle without evidence of significant treatment-related toxicity or clinically significant progressive disease will continue to receive treatment for up to six cycles.

SUMMARY:
The primary objective of this study is to determine the maximum tolerated dose, dose limiting toxicity, safety and tolerability of TH-302 in patients with acute leukemias, advanced phase chronic myelogenous leukemia (CML), high risk myelodysplastic syndromes, advanced myelofibrosis or relapsed/refractory chronic lymphocytic leukemia (CLL).

DETAILED DESCRIPTION:
Tumor hypoxia has been associated with resistance to chemotherapy and radiotherapy (Brown et al, 2004; Boyle 2006). TH-302, a hypoxia activated prodrug (HAP), exploits the hypoxic nature of tumors while having little or no effect on normal tissue. TH-302 belongs to a class of alkylating agents called oxazaphosphorines which have major experimental and clinical activity (Brock 1989). Since TH-302 is selectively targeted to the hypoxic microenvironment, this agent may represent an improvement over other agents in this class. Preclinical data support the hypothesis that TH-302 targets hypoxic regions of tumors and also is able to kill other tumor cells in normoxic regions as a result of cytotoxin diffusion, leading to significant effects on tumor growth. Preclinical data has shown that TH-302 has anti-tumor activity in multiple myeloma cells in vivo and in vitro.

Additional preclinical data demonstrated the marked expansion of the hypoxic bone marrow areas in diseased mice with ALL. These results suggest that this agent may be useful in treating advanced leukemias. The drug is stable in plasma and liver, does not appear to be at risk for drug-drug interactions, and has mild, reversible toxicities. In this dose-escalation study, patients with advanced leukemias will receive infusions of TH-302 to determine the maximum tolerated dose.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Ability to understand the purposes and risks of the study and has signed a written informed consent form approved by the investigator's IRB/Ethics Committee.
* Relapsed/refractory leukemias for which no standard therapy options are anticipated to result in a durable remission.
* Acute myelogenous leukemia (AML) by WHO classification relapsed or refractory to standard chemotherapy; unsuitable for standard chemotherapy or unwilling to undergo standard chemotherapy.
* Acute lymphoblastic leukemia (ALL) relapsed or refractory to standard chemotherapy; unsuitable for standard chemotherapy or unwilling to undergo standard chemotherapy. Philadelphia chromosome (Ph) positive ALL eligible if failed prior tyrosinekinase inhibitor therapy.
* Chronic myelogenous leukemia (CML) in accelerated or blast phase failing prior tyrosine kinase-containing therapy
* High-risk myelodysplastic syndrome (MDS) [i.e. refractory anemia with excess blasts (RAEB-1 or RAEB-2) by WHO classification] or chronic myelomonocytic leukemia (CMML) with >5% marrow blasts, relapsed or refractory to standard therapy
* Chronic lymphocytic leukemia (CLL) relapsed or refractory to standard therapy, not eligible for protocols of higher priority
* Advanced myelofibrosis (MF) resistant or refractory to standard therapy; or untreated with one of following features (1) hemoglobin < 10 g/dL, (2) platelet count < 100 x 109/L, WBC < 4 or > 30 x 109/L, or splenomegaly ≥ 10 cm below left costal margin
* Age > 60 years with AML not candidates for or have refused standard chemotherapy, excluding subjects with acute promyelocytic leukemia (APL) or with favorable cytogenetic abnormalities [inv16, t(8;21)].
* ECOG performance status of less than or equal to 3
* Adequate organ function as indicated by the following laboratory assessments performed within 14 days prior to the first dose of study drug:
* Total bilirubin ≤ 1.5 times upper limit of normal (x ULN) (≤ 3 x ULN if due to leukemic involvement or Gilbert's syndrome).
* Aspartate aminotransferase or alanine aminotransferase ≤ 2.5 x ULN (≤ 5.0 x ULN if due to leukemic involvement)
* Serum creatinine ≤ 1.5 x ULN.
* All women of childbearing potential must have a negative serum pregnancy test and women and men subjects must agree to use effective means of contraception (surgical sterilization or the use or barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel or an IUD) with their partner from entry into the study through 6 months after the last dose

Exclusion Criteria:

* New York Heart Association (NYHA) Class III or IV, cardiac disease, myocardial infarction within 6 months prior to Day 1, or unstable arrhythmia
* Seizure disorders requiring anticonvulsant therapy
* Severe chronic obstructive pulmonary disease with hypoxemia or in the opinion of the investigator any physiological state leading to hypoxemia
* Major surgery, other than diagnostic surgery, within 4 weeks prior to Day 1, without complete recovery
* Active uncontrolled infection
* Systemic chemotherapy (with the exception of hydroxyurea and/or steroids) within 14 days (or within 5 half-lives for an investigational agent) prior to first dose of study drug, unless there is evidence of rapidly progressive disease. Concurrent therapy for CNS prophylaxis or continuation of therapy for controlled CNS disease is permitted.
* Known active infection with HIV, hepatitis B, or hepatitis C
* Patients who have exhibited allergic reactions to a similar structural compound, biological agent, or formulation (containing solutol and/or propylene glycol)
* Females who are pregnant or breast-feeding
* Concomitant disease or condition that could interfere with the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study
* Unwillingness or inability to comply with the study protocol for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-06; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose of TH-302 | 2 years
To determine the dose-limiting toxicity of TH-302 | 2 years
TO determine the number of participants with Adverse Events as a measure of safety and tolerability | 2 years

SECONDARY OUTCOMES:
To determine the efficacy of TH-302 via specific response criteria | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Marina Konopleva, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas M.D. Anderson Cancer Center, Houston, Texas, United States